CLINICAL TRIAL: NCT01162733
Title: A Randomized Prospective Study of Vancomycin Dosing in the Emergency Department: Will a Loading Dose of 30mg/kg Lead to a More Rapid Attainment of Therapeutic Levels?
Brief Title: Loading Vancomycin Doses in the Emergency Department
Acronym: Loaded
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30029
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Results first posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Infectious Disease
Keywords: Vancomycin; Therapeutic Levels; Infectious Disease; Recommendations
MeSH Terms: conditions — Communicable Diseases | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Drug 1 (Active Comparator): Vancomycin 15mg/kg
  Interventions: Drug: Vancomycin
- Study Drug 2 (Active Comparator): Vancomycin 30mg/kg
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — 15mg/kg
  Arms: Study Drug 1
Drug: Vancomycin — 30mg/kg
  Arms: Study Drug 2

SUMMARY:
In 2008, our ED administered an average of 245 doses of vancomycin per month. Currently there is no consistency in the ED practice in regards to vancomycin dosing. In 2009, the IDSA put forth new recommendations for vancomycin dosing in order to achieve therapeutic levels more rapidly. It has been hypothesized that if therapeutic levels are reached more rapidly then patients will in turn have better clinical outcomes and that the development of resistant organisms will be decreased. Methicillin resistant Staphylococcus aureus (MRSA) has emerged as one of the most deadly pathogens that are currently plaguing our patient population. Vancomycin is one of only a few antibiotics that are effective for treating MRSA. It is imperative that the ED physicians consistently and correctly dose vancomycin in order to give the patients the best chance to fight infection while helping to prevent further resistance in this already highly resistant organism. It is believed this study will reveal that the new dosing recommendations by the IDSA will lead to the achievement of therapeutic levels more rapidly. This information will in turn help to convince ED physicians that a change in current clinical practice is warranted and ultimately lead to better clinically outcomes for the patients.

DETAILED DESCRIPTION:
Recently, the Infectious Disease Society of America (IDSA) has released new dosing recommendations for intravenous (IV) vancomycin. These new recommendations suggest administering an initial dose of 25-30 mg/kg of vancomycin as opposed to 10-15 mg/kg which is more traditionally done. Currently in the Emergency Department (ED) some practitioners are using the new IDSA dosing recommendations for vancomycin, while other practitioners have not changed their clinical practice. There is currently little data available to suggest that implementing these new vancomycin dosing regimens in the ED will achieve therapeutic vancomycin levels more rapidly than our traditional dosing practice.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Treated in Christiana Emergency Department
* Receiving Vancomycin for an infection or presumed infection
* Being admitted to Christiana Hospital
* Planned continued use of Vancomycin after admission.

Exclusion Criteria:

* Less than 18 years of age
* Weight greater than 120 kg.
* Concurrent use of aminoglycosides or acyclovir
* Sepsis patients being admitted to ICU with presumed diagnosis of pneumonia
* Patients currently undergoing dialysis
* Pregnant or breast feeding
* No plan to continue Vancomycin after admission.
* Creatinine clearance less than 50ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Levine, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Chrisitana Care Health System-Christiana Hospital, Newark, Delaware, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Drug 1: Vancomycin 15mg/kg
  Vancomycin : 15mg/kg
- Study Drug 2: Vancomycin 30mg/kg
  Vancomycin : 30mg/kg
Period: Overall Study
Arm/Group | Study Drug 1 | Study Drug 2
Started | 49 | 50
Completed | 22 | 25
Not Completed | 27 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Drug 1 | Study Drug 2 | Total
Number analyzed (Participants) | 49 | 50 | 99
Age, Customized [Number; unit: participants]
  Greater than 18 years of age | 49 | 50 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 25 | 28 | 53
Region of Enrollment [Number; unit: participants]
  United States | 49 | 50 | 99

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants First Achieving Therapeutic Levels at 36 Hours
Description: The objective is to determine if therapeutic levels were reached more rapidly with the implementation of an initial vancomycin loading dose of 30 mg/kg as compared to 15mg/kg.
Time Frame: 36 hours
Measure: Number; unit: percentage of participants
Arm/Group | Study Drug 1 | Study Drug 2
Number analyzed (Participants) | 49 | 50
percentage of participants | 20 | 18

2. Primary Outcome: Percentage of Participants First Achieving Therapeutic Levels at 12 Hours
Description: Percentage of patients reaching a therapeutic level defined as greater than 15 mcg/mL
Time Frame: 12 hours
Measure: Number; unit: percentage of participants
Arm/Group | Study Drug 1 | Study Drug 2
Number analyzed (Participants) | 49 | 50
percentage of participants | 3 | 34

ADVERSE EVENTS:
Arm/Group | Study Drug 1 | Study Drug 2
Serious Adverse Events (participants affected / at risk) | 0/49 | 2/50
Other Adverse Events (participants affected / at risk) | 3/49 | 3/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug 1 (N=49) | Study Drug 2 (N=50)
New onset Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Drug 1 (N=49) | Study Drug 2 (N=50)
Allergic Reaction (Immune system disorders) | 2 (2) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No